CLINICAL TRIAL: NCT01279694
Title: Phase I/II Trial of Carfilzomib Plus Melphalan and Prednisone in Elderly Untreated Patients With Multiple Myeloma.
Brief Title: Trial of Carfilzomib Plus Melphalan and Prednisone in Elderly Untreated Patients With Multiple Myeloma (CARMYSAP)
Acronym: CARMYSAP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10/3-D
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2013-09

CONDITIONS: Myeloma
Keywords: newly-diagnosed multiple myeloma.
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — carfilzomib; Melphalan; Prednisone

INTERVENTIONS:
Drug: Carfilzomib — There are 9 cycle of 20mg/m²,Intravenous for J1, J2, J8, J9, J22, J23, J29 and 30 days with 12 days rest (42 day cycle) for the first cohort; or 20mg/m²,Intravenous for J1, J2, and 27 mg/m² for J8, J9, J22, J23, J29 and 30 days with 12 days rest (42 day cycle) for the second cohort for the last, third cohort 20mg/m²,Intravenous for J1, J2, and 36 mg/m² for J8, J9, J22, J23, J29 and 30 days with 12 days rest (42 day cycle)and the fourth cohort 20mg/m²,Intravenous for J1, J2, and 45 mg/m² for J8, J9, J22, J23, J29 and 30 days with 12 days rest (42 day cycle). .
Drug: Melphalan — from 9 cycle: 9 mg/m²/day PO from day 1-4
  Other Names: alkéran
Drug: Prednisone — from 9 cycle: 60 mg/m²/day PO from day 1-4

SUMMARY:
Phase I/II trial of Carfilzomib plus melphalan and prednisone in elderly untreated patients with multiple myeloma. Nine: University Hospital of Nantes, University Hospital of Nancy, University Hospital of Lille, University Hospital of Tours, department Hospital of La Roche Sur Yon, University Hospital of Reims, University Hospital of Clermont-Ferrand, University Hospital of Toulouse, University Hospital of Dijon Newly diagnosed symptomatic Multiple Myeloma > 65 years. Treatment comprises an initial phase consisting of nine 6-week cycles of Carfilzomib on Days 1, 2, 8, 9, 22, 23, 29, 30 (carfilzomib is administered at 20 mg/m2 on Days 1 and 2 of the first cycle and 20, 27, 36 or 45 mg/m2 thereafter) followed by a 12 day rest period (42-day cycle), in combination with oral Melphalan 9 mg/m² and oral prednisone 60mg/m², both on days 1 to 4.

Phase I: Identification of Maximum Tolerated Dose (MTD)

Carfilzomib will be administered at a dose of 20mg/m² for all doses to the first cohort of 6 patients. If dose-limiting toxicities (DLTs) occurred in fewer than 2 of these patients, the next cohort of 6 patients (cohort 2) will receive a dose of 20/27 mg/m² where the 20 mg/m² dose is administered on Day 1 and 2 of Cycle 1 only and then 27 mg/m² for all subsequent doses. If DLTs occurred in fewer than 2 of the patients in cohort 2, the third cohort of 6 patients will receive a dose of 20/36 mg/m² where the 20 mg/m² dose is administered on Day 1 and 2 of Cycle 1 only and then 36 mg/m² for all subsequent doses. If DLTs occurred in fewer than 3 of the patients in cohort 3 the fourth cohort of 6 patients will receive a dose of 20/45 mg/m² where the 20 mg/m² dose is administered on Day 1 and 2 of Cycle 1 only and then 45 mg/m² for all subsequent doses. If at any time during cycle 1 of a dose cohort, ≥ 2 subjects experience a drug-related DLT, the MTD will have been exceeded, additional enrollment within the cohort will cease, and dose escalation will stop. The MTD will be defined as the dose level below which DLT is observed in ≥ 33% (i.e. ≥ 2 of 6) subjects in a cohort. The following are defined as DLTs:

* Any hematologic toxicity of grade 4 intensity or preventing administration of 2 or more of the 8 carfilzomib doses of the first treatment cycle except a) grade 4 thrombocytopenia without bleeding lasting ≤ 7 days or b) grade 4 neutropenia lasting ≤ 7 days
* Grade ≥ 3 febrile neutropenia
* Grade ≥ 3 gastrointestinal toxicities (except for grade ≥ 3 nausea/ vomiting if the patient had not received adequate antiemetic prophylaxis)
* Any other grade ≥ 3 nonhematologic toxicity considered related to CMP by the principal investigator.
* Grade ≥ 3 peripheral neuropathy persisting for more than 3 weeks after discontinuation of study drugs.

Adverse events (AEs) will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE, version 4.0). MTD determination will be based on occurrence of DLTs during the first induction treatment cycle only.

Phase II: Expanded Cohort. After identification of the MTD, it is planned for the dose cohort to be expanded to include up to a total of 20 patients treated at the MTD for the phase II part of the study. A full treatment course is the same as for phase I: nine 6-week cycles of CMP.

PRIMARY ENDPOINT Phase I: MTD of combination Phase II: Overall response rate [(ORR), consisting of complete response (CR), very good partial response (VGPR), and partial response (PR) SECONDARY ENDPOINTS Safety and tolerability of CMP Clinical benefit response [(CBR = ORR + minimal response (MR)], Progression-free survival (PFS), Duration of response Overall survival (OS). Safety data analysis will be conducted on all subjects receiving at least one dose of study treatment. Analyses will consist of data summaries for reported AEs. The number and percentage of subjects experiencing one or more AEs will be summarized by dose, relationship to study drugs, and severity. AEs will be coded using MedDRA terminology.

Disease Response Analyses: Overall response rate (ORR = CR + VGPR + PR) to treatment will be measured using the International Myeloma Working Group (IMWG) criteria. Clinical benefit response (CBR = ORR + MR) will be determined using minimal response (at least 6 weeks duration) as defined by the European Group for Blood and Marrow Transplant (EBMT). The distribution of subjects by response category will be made overall and by dose cohort. Time-to-event endpoints will be evaluated with the use of the Kaplan-Meier method and plots will be provided. Analysis of time-to-event outcomes will be performed for the overall sample.

DETAILED DESCRIPTION:
The primary objectives of this phase I/II study are to identify the most appropriate dose of Carfilzomib in combination with a standard MP treatment regimen (phase I) and to evaluate the efficacy of Carfilzomib plus MP (CMP) in terms of overall response rate [(ORR), consisting of complete response (CR), very good partial response (VGPR), and partial response (PR) (phase II)]. Phase I/II single arm open label

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance status (KPS) of at least 60%
* Life expectancy of more than 3 months.
* Must understand and voluntarily sign an informed consent form
* Age >65 years at the time of signing consent
* Previously untreated, symptomatic multiple myeloma as defined by the 2 criteria below:○ MM diagnostic criteria (all 3 required):· Monoclonal plasma cells in the bone marrow ≥10% and/or presence of a biopsy-proven plasmacytoma· Monoclonal protein present in the serum and/or urine· Myeloma-related organ dysfunction (at least 1 of the following) [C] Calcium elevation in the blood (serum calcium >10.5 mg/L or upper limit of normal)[R] Renal insufficiency (serum creatinine > 2 mg/dL)[A] Anemia (hemoglobin <10 g/dL or 2 g < normal)[B] Lytic bone lesions or osteoporosisAND have measurable disease by protein electrophoresis analyses as defined by one or more of the following:· IgG multiple myeloma: Serum monoclonal paraprotein (M protein) level by SPEP ³ 0.5 g/dL or urine M-protein level ³ 200 mg/24 hours· IgA multiple myeloma: Serum M-protein level ³ 0.5 mg/dL or urine M-protein level ³ 200 mg/24 hours· IgM multiple myeloma (IgM M-protein plus lytic bone disease documented by skeletal survey plain films): Serum M-protein level ≥ 1.0 g/dL or urine M-protein level ≥ 200 mg/24 hours· IgD multiple myeloma: Serum M-protein level ³ 0.05 g/dL or urine M-protein level ³ 200 mg/24 hours Light chain multiple myeloma: Patients with serum free light chain disease in whom the involved light chain measures ≥ 10 mg/dL
* ECOG performance status of 0, 1, or 2
* Able to adhere to the study visit schedule and other protocol requirements
* Affiliation number to National Health Care System

Exclusion Criteria:

* Patients are ineligible if they meet any of the following criteria: 1 Previous treatment with antimyeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid [i.e., less than or equal to the equivalent of dexamethasone 40 mg/day for 4 days; such a short course of steroid treatment must not have been given within 28 days (4 weeks) of consent]).
* Any serious medical condition that places the patient at an unacceptable risk if he or she participates in this study.
* Female of childbearing potential
* Any of the following laboratory abnormalities:· Absolute neutrophil count (ANC) < 1,000 cells/mL (1.0 × 109/L) · Platelet count < 50,000 cells/mL (50 × 109/L) for patients in whom < 50% of bone marrow nucleated cells are plasma cells; but platelet count <30,000 cells/mL for patients in whom ³ 50% of bone marrow nucleated cells are plasma cells · Serum SGPT/ALT > 3.0 × upper limit of normal (ULN); Bilirubin >2 × ULN [ALT more specific to liver]· Creatinine clearance ≤ 30 mL/min (Cockcroft-Gault calculation)5 Prior history of malignancies, other than multiple myeloma, unless the subject has been free of the disease for ³ 3 years. Exceptions include the following:o Basal cell carcinoma of the skin Squamous cell carcinoma of the skin Carcinoma in situ of the cervix Carcinoma in situ of the breast6 Incidental histological finding of prostate cancer (TNM stage of T1a or T1b) Peripheral neuropathy of > grade 2 severity.
* Known HIV positivity or active infectious hepatitis, type A, B, or C.
* Myocardial infarction within 3 months of enrollment, unstable angina within 2 months or New York Heart Association class III or IV heart failure.
* Oral or IV fluid hydration contraindicated

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Phase I: determination of MTD by evaluation of hematological and non hematological toxicity

SECONDARY OUTCOMES:
Safety of CMP Clinical benefit response [(CBR = ORR + minimal response (MR)], Progression-free survival (PFS), Duration of response Overall survival (OS).
Tolerability of CMP Clinical benefit response [(CBR = ORR + minimal response (MR)], Progression-free survival (PFS), Duration of response Overall survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Moreau, Principal Investigator — Nantes University Hospital; Carine Chaleteix, Principal Investigator — University Hospital, Clermont-Ferrand; Denis Caillot, Principal Investigator — CH DIJON; Thierry FACON, Principal Investigator — CHRU - Hôpital Claude Huriez Lille; Cyril Hulin, Principal Investigator — Hôpital de Brabois Nancy; Brigitte Kolb, Principal Investigator — Hôpital R. Debré Reims; Hervé Maisonneuve, Principal Investigator — CHD La Roche sur Yon; Michel Attal, Principal Investigator — CHRU - Hôpital Purpan Toulouse; Benboubker, Principal Investigator — CHRU - Hôpital Bretonneau Tours
Locations (1):
- CHU de Nantes, Nantes, France

REFERENCES:
- [Derived] Moreau P, Kolb B, Attal M, Caillot D, Benboubker L, Tiab M, Touzeau C, Leleu X, Roussel M, Chaleteix C, Planche L, Chiffoleau A, Fortin J, Avet-Loiseau H, Mary JY, Hulin C, Facon T. Phase 1/2 study of carfilzomib plus melphalan and prednisone in patients aged over 65 years with newly diagnosed multiple myeloma. Blood. 2015 May 14;125(20):3100-4. doi: 10.1182/blood-2015-02-626168. Epub 2015 Mar 17. PMID 25784682